CLINICAL TRIAL: NCT04838899
Title: Stereotactic Ablative Radiotherapy for Oligoprogressive Metastatic Castration-Resistant Prostate Cancer During Abiraterone Therapy
Brief Title: Stereotactic Ablative Radiation Therapy for Abiraterone-Resistant, Oligoprogressive Metastatic Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Urban Emmenegger, Medical Oncologist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #351
Record Dates: First submitted 2021-04-03; First posted 2021-04-09 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Oligoprogressive; Castration-Resistant Prostate Cancer
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): All metastases that fulfill the definition of oligoprogression seen on conventional imaging will be treated with standard SABR dose fractionation schemes routinely used at Sunnybrook Odette Cancer Centre. The prostate (if present and not previously treated) will be treated to a dose of 35 Gy in 5 fractions. Non-spine bone metastases will be treated to a dose of 30-40 Gy in 5 fractions. Spine metastases will be treated to a dose of 24 Gy in 2-3 fractions or 30-40 Gy in 5 fractions. Involved lymphadenopathy will be treated to a dose of 30-40 Gy in 5 fractions. Similarly, brain, lung, liver, and adrenal metastases will be treated with standard Sunnybrook SABR doses. Patients will remain on abiraterone during and after SABR treatments.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SABR)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SABR) — SABR to oligoprogressive metastases while continuing abiraterone therapy

SUMMARY:
There is increasing worldwide interest in exploring stereotactic ablative body radiotherapy (SABR) for treating metastases in men with prostate cancer, including for the treatment of oligoprogressive metastases. The latter applies to a situation whereby patients with widespread metastases undergoing systemic therapy present with a solitary or a few metastatic tumors that progress, while all other metastases are stable or responding. The usual practice would be to change systemic therapy at this point, but another approach is to locally ablate the "rogue" metastases and continue the same systemic therapy. SABR used in this scenario may delay the need to switch to another line of systemic therapy and improve progression-free survival while patients stay on the same systemic therapy.

DETAILED DESCRIPTION:
There is increasing worldwide interest in exploring the use of SABR for metastatic, treatment-naive prostate cancer, eg for delaying the need to start androgen deprivation therapy (ADT), and ultimately to improve patient outcome.

Another potential use of SABR for metastatic prostate cancer is in the setting of oligoprogression. In patients undergoing systemic therapy, oligoprogression describes the clinical situation where a solitary or a few metastatic tumors progress, while all other metastases are stable or responding. The usual practice would be to change systemic therapy at this point, but another approach is to locally ablate the "rogue" metastases and continue the same systemic therapy. There is limited clinical evidence for such an approach, eg in renal cell and non-small cell lung cancer.

While there is a lack of published evidence of such an approach in metastatic castration-resistant prostate cancer (mCPRC), SABR for oligoprogressive mCRPC in men undergoing abiraterone therapy may delay the need to switch to another line of systemic therapy, such as chemotherapy, and thereby to improve progression-free survival while patients stay on the same systemic therapy.

mCRPC is a unique solid tumor to study the oligoprogressive setting for several reasons. First, there still remains a limited number of proven systemic agents in the CRPC setting. Second, serum prostate specific antigen (PSA) is an excellent biomarker of prostate cancer activity, which is easy to collect and analyze to monitor treatment response and disease progression. Third, because of the low α/β value of prostate cancer, hypofractionated SABR may be a very effective and convenient way to eradicate areas of known disease.

The primary objective of this phase I study is to determine the incidence of acute and late toxicities associated with delivering SABR to all progressive metastatic sites in patients with metastatic CRPC who present with oligoprogression while on abiraterone. We also aim to obtain preliminary efficacy data of this novel approach. Patients will remain on abiraterone after SABR to measure the added progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0-1.
* Histologic confirmation of prostate adenocarcinoma.
* Documentation of metastatic, castration-resistant prostate cancer.
* Patient being treated with abiraterone.
* Evidence of oligoprogression (according to RECIST [V1.1] and/or Prostate Cancer Working Group criteria [PCWG3], as applicable), applying any of the following: (i) ≤ 5 metastatic lesions progressing on conventional imaging (≤ 3 progressing metastases in any one organ system) while all other metastases are controlled or responding; (ii) PSA progression only, but in the setting of oligometastases (≤ 5 metastatic lesions seen on imaging, with ≤ 3 metastases in any one organ system); in this setting, all metastases will be irradiated.
* All metastases of interest amenable to SABR.

Exclusion Criteria:

* Patients presenting with unequivocal clinical progression, defined as one of the following: (i) cancer pain requiring the initiation of opioid therapy; (ii) immediate need for cytotoxic chemotherapy as per treating physician's discretion; or (iii) deterioration of performance status to grade ≥ 3 according to ECOG.
* Evidence of spinal cord compression.
* Prior malignancy within the past 5 years, excluding non-melanoma skin cancer, and in-situ cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-07-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
SABR-related toxicities | 12 months
  Incidence of acute and late toxicities (including radiation induced bone fractures) after comprehensive SABR to all progressing metastases seen on conventional imaging.
Progression-free survival | 24 months
  Time to clinical (i.e., radiological and/or symptomatic) progression following SABR.

SECONDARY OUTCOMES:
Biochemical progression-free survival | 24 months
  Time to PSA progression
Time to changing systemic therapy | 24 months
  Time to starting subsequent line of systemic therapy
Radiographic local control rate of the SABR-treated areas | 24 months
  Monitoring lack of progression of oligoprogressive sites of disease
Radiographic distant progression-free survival | 24 months
  Time to metastatic progression outside of SABR-treated areas
Overall survival | 36 months
  Time to death from prostate cancer or other cause
Quality of Life (QoL) assessment | 12 months
  QoL assessment using EORTC QLQ-C30 at baseline, plus 1, 3, 6, 9 and 12 months after SABR

CONTACTS AND LOCATIONS:
Locations (1):
- Odette Cancer Centre, Toronto, Ontario, Canada